CLINICAL TRIAL: NCT06595836
Title: Evaluation of the Performance and Acceptability of a Synthetic Polyisoprene Male Condom Compared to a Natural Rubber Latex Condom (Phase II Slippage/Breakage Study)
Brief Title: Evaluation of the Performance and Acceptability of a Synthetic Polyisoprene Male Condom Compared to a Natural Rubber Latex Condom
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Nippon Rubber Industry Public Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TNR-01
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Condom Use

STUDY DESIGN:
Intervention Model Description: This study is a masked (investigators, research staff), two-way crossover, randomized to sequence of use study designed to evaluate the acceptability and functional performance (breakage, slippage) of a silicone lubricated polyisoprene condom and a silicone lubricated natural rubber latex condom
Who Masked: Investigator, Outcomes Assessor
Masking Description: Each product will be labeled with a randomly generated code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- polyisoprene condoms lubricated with a silicone lubricant (Experimental): polyisoprene condoms lubricated with a silicone lubricant
  Interventions: Device: Silicone Lubricated Synthetic polyisoprine condom
- commercial latex condoms with a silicone lubricant (Active Comparator): commercial latex condoms with a silicone lubricant
  Interventions: Device: Silicone Lubricated Natural Rubber Latex Condom

INTERVENTIONS:
Device: Silicone Lubricated Synthetic polyisoprine condom — Synthetic polyisoprene condom are made from softer materials for a more natural feel and increased sensitivity
  Arms: polyisoprene condoms lubricated with a silicone lubricant
Device: Silicone Lubricated Natural Rubber Latex Condom — Natural rubber latex condoms are made from natural rubber
  Arms: commercial latex condoms with a silicone lubricant

SUMMARY:
This study is a masked (investigators, research staff), two-way crossover, randomized to sequence of use study designed to evaluate the acceptability and functional performance (breakage, slippage) of a silicone lubricated polyisoprene condom and a silicone lubricated natural rubber latex condom.

DETAILED DESCRIPTION:
Three hundred (300) couples will be enrolled and asked to use five condoms of each of the two types of lubricated condoms to yield a potential sample size of 1500 uses for each type of lubricated condom. To minimize a potential learning effect, couples will be randomly assigned to the sequence of use of each type of lubricated condom.

The primary objective of this study is to examine the slippage, breakage and acceptability of a new polyisoprene male condom compared to a natural rubber latex condom. The study will assess safety in terms of adverse events and user acceptability will be evaluated by comparing physical attributes of the polyisoprene and latex control condoms, as well as perceptions about using the devices.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 45 (inclusive)
2. Willing and able to give written or electronic informed consent
3. Willing to respond to questions concerning their reproductive and contraceptive history and use of condoms contained either on self-administered questionnaires or interviews
4. Be sexually active (defined as averaging one vaginal coital act per week)
5. Protected against pregnancy by oral contraceptives, an IUD, an implant, contraceptive injections, contraceptive patch, or sterilization (tubal ligation or vasectomy)
6. Willing to use the study products for ten acts of vaginal intercourse within six weeks of study entry
7. In a mutually monogamous relationship with their study partner for at least 3 months and be willing to remain mutually monogamous throughout study participation
8. Agree not to use any vaginal or sexual lubricant except the product supplied by the study
9. Agree not to wear any genital piercing jewelry while using the study condoms
10. Agree not to use sex toys or drugs intended to enhance or diminish sexual response when using study condoms
11. Agree to return any unopened condoms
12. Reachable by telephone
13. Has home internet access, a valid personal email for each partner, reachable by phone, ability to videoconference and use electronic consent technology
14. Male partner agrees to ejaculate during vaginal intercourse
15. Willing to provide photo identification-

Exclusion Criteria:

1. Currently participating in another similar clinical study or employed by a condom manufacturer or Essential Access Health
2. Female partner self-reported as pregnant
3. Allergic to natural rubber latex or polyisoprene, or has a history of recurrent adverse events following use of latex or polyisoprene products
4. Unable to follow instructions or strictly adhere to the visit schedule
5. At significant (high) risk of sexually transmitted infections, including HIV infection, or having a medical history of recurrent, serious sexually transmitted infection (e.g. gonorrhea, syphilis, Chlamydia)
6. Currently using condoms for protection against a known sexually transmitted infection
7. Taking any internally applied medication or oral medication to treat a genital condition
8. Male partner has had difficulty achieving or maintaining an erection, or achieving ejaculation in the last month under typical circumstances/ conditions.
9. Any self-reported genital condition (e.g. itching, burning, irritation, etc.) which, in the opinion of the investigator, could affect use of the study condoms or the ability to interpret study data -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Total Clinical Failure | 5 -7 weeks
  The total clinical failure rate is defined as the number of condoms that broke or slipped completely off the penis during intercourse or withdrawal over the number of condoms used for vaginal intercourse.

SECONDARY OUTCOMES:
Clinical Breakage | 5 - 7 weeks
  The clinical breakage rate is defined as the number of condoms that broke during intercourse or withdrawal over the number of condoms used for vaginal intercourse.
Clinical Complete Slippage | 5-7 weeks
  The clinical complete slippage rate is defined as the number of condoms that slipped completely off the penis during intercourse or withdrawal over the number of condoms used for vaginal intercourse

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Essential Access, Berkeley, California
  - Essential Access, Los Angeles, California